CLINICAL TRIAL: NCT02519348
Title: A Study of Safety, Tolerability, and Clinical Activity of Durvalumab and Tremelimumab Administered as Monotherapy, or Durvalumab in Combination With Tremelimumab or Bevacizumab in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Durvalumab or Tremelimumab Monotherapy, or Durvalumab in Combination With Tremelimumab or Bevacizumab in Advanced Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00022; 2024-517085-41-00 (Registry Identifier: CTIS); 2015-001663-39 (EudraCT Number)
Record Dates: First submitted 2015-07-30; First posted 2015-08-10 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Immunotherapy; Antibodies, Monoclonal; Tremelimumab; MEDI4736; Durvalumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tremelimumab; durvalumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg (Experimental): Participants in Part 1A (safety run-in cohort) and Part 1 B (efficacy-gating cohort) will receive tremelimumab 1 mg/kg every 4 weeks (Q4W) 4 doses and durvalumab 20 mg/kg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Biological: Tremelimumab; Biological: Durvalumab
- Parts 2 and 3: Durvalumab 1500 mg (Experimental): Participants will receive durvalumab 1500 mg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Biological: Durvalumab
- Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg (Experimental): Participants will receive tremelimumab 300 mg 1 dose and durvalumab 1500 mg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Biological: Tremelimumab; Biological: Durvalumab
- Parts 2 and 3: Tremelimumab 750 mg (Experimental): Participants will receive tremelimumab 750 mg Q4W 7 doses followed by every 12 weeks (Q12W) until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Biological: Tremelimumab
- Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg (Experimental): Participants will receive tremelimumab 75 mg Q4W 4 doses and durvalumab 1500 mg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first. Participant recruitment to this arm was closed following protocol amendment 5.
  Interventions: Biological: Tremelimumab; Biological: Durvalumab
- Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg (Experimental): Participants will receive durvalumab 1120 mg and bevacizumab 15 mg/kg every 3 weeks (Q3W) until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first
  Interventions: Biological: Durvalumab; Biological: Bevacizumab
- China Cohort: Durvalumab 20 mg/kg (Experimental): Participants will receive durvalumab 20 mg/kg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Biological: Durvalumab
- China Cohort: Tremelimumab 10 mg/kg (Experimental): Participants will receive tremelimumab 10 mg/kg Q4W 7 doses followed by Q12W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Biological: Tremelimumab
- China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg (Experimental): Participants will receive tremelimumab 1 mg/kg Q4W 4 doses and durvalumab 20 mg/kg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Biological: Tremelimumab; Biological: Durvalumab

INTERVENTIONS:
Biological: Tremelimumab — Tremelimumab will be administered by IV infusion according to doses and frequency mentioned in arms' description.
  Arms: China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg; China Cohort: Tremelimumab 10 mg/kg; Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg; Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg; Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg; Parts 2 and 3: Tremelimumab 750 mg
Biological: Durvalumab — Durvalumab will be administered by IV infusion according to doses and frequency mentioned in arms' description.
  Other Names: MEDI4736
  Arms: China Cohort: Durvalumab 20 mg/kg; China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg; Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg; Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg; Parts 2 and 3: Durvalumab 1500 mg; Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg; Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg
Biological: Bevacizumab — Bevacizumab 15 mg/kg will be administered by IV infusion every 3 weeks until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
  Arms: Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg

SUMMARY:
This is a multicenter, open-label, stratified, randomized study to evaluate the safety, tolerability, antitumor activity, pharmacokinetics, pharmacodynamics, and immunogenicity of durvalumab or tremelimumab monotherapy, or durvalumab in combination with tremelimumab or bevacizumab in advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
The study will comprise of 6 parts. Participants in Part 1A (safety run-in cohort), Part 1B (efficacy-gating cohort), Part 2A, and Part 4 will receive weight-based dosing regimens; and participants in Part 2B and Part 3 will receive fixed dosing regimens. Part 1A Stage 2 of the study may start after the first 3 participants in Stage 1 have been observed on study for at least 4 weeks. In addition, a separate cohort of participants will be enrolled in mainland China (China cohort) once global recruitment in Part 2A will be closed.

* In Part 1 (both 1A and 1B), participants will receive tremelimumab 1 mg/kg intravenous (IV) every 4 weeks (Q4W) 4 doses and durvalumab 20 mg/kg Q4W.
* In Part 2A, participants will be randomized in a 1:1:1 ratio to receive:

  * Durvalumab 20 mg/kg Q4W
  * Tremelimumab 10 mg/kg Q4W × 7 doses followed by every 12 weeks (Q12W)
  * Tremelimumab 1 mg/kg Q4W × 4 doses + durvalumab 20 mg/kg Q4W, followed by durvalumab 20 mg/kg Q4W
* In China cohort, Part 2A study design will be followed.
* In Part 2B, participants will receive tremelimumab 300 mg × 1 dose + durvalumab 1500 mg Q4W.
* In Part 3, participants will be randomized in a 2:2:1:2 ratio to receive:

  * Durvalumab 1500 mg Q4W
  * Tremelimumab 300 mg × 1 dose + durvalumab 1500 mg Q4W
  * Tremelimumab 750 mg Q4W for 7 doses followed by Q12W
  * Tremelimumab 75 mg Q4W × 4 doses + durvalumab 1500 mg Q4W, followed by durvalumab 1500 mg Q4W.

Following protocol amendment 5, enrollment into 'Tremelimumab 75 mg Q4W × 4 doses + durvalumab 1500 mg' arm will close. Participants will be randomized at a ratio of 2:1:2 in 'Durvalumab 1500 mg Q4W', 'Tremelimumab 750 mg Q4W for 7 doses followed by Q12W', and 'Tremelimumab 300 mg × 1 dose + durvalumab 1500 mg Q4W' arms, respectively.

• In Part 4, participants will receive durvalumab 1120 mg (15 mg/kg) + bevacizumab 15 mg/kg every 3 weeks (Q3W).

Participants will receive the treatment until confirm progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurs first.

All participants will be followed for survival until the end of study visit (last participant discontinues the study treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants
2. 18 years and older (Japan-20 years and older)
3. Confirmed hepatocellular carcinoma (HCC) based on histopathological findings from tumor tissues. Advanced HCC with diagnosis confirmed pathologically or with noninvasive methods.
4. Immunotherapy-naïve
5. Have either progressed on, are intolerant to, or refused treatment with sorafenib or another approved TKI. For arm 5 only: Have not received any prior systemic therapy for HCC.

Exclusion Criteria:

1. Prior exposure to immune-mediated therapy
2. Hepatic encephalopathy within past 12 months or requirement for medications to prevent or control encephalopathy
3. Gastrointestinal bleeding (eg, esophageal varices or ulcer bleeding) within 12 months
4. Ascites requiring non-pharmacologic intervention (eg, paracentesis) to maintain symptomatic control, within 6 months prior to the first scheduled dose.
5. Main portal vein thrombosis (Vp4) as documented on imaging
6. Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment
7. Active or prior documented autoimmune or inflammatory disease with some exceptions
8. Current or prior use of immunosuppressive medication within 14 days with some exceptions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2026-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune, LLC MedImmune, LLC, Study Director — MedImmune LLC
Locations (38):
- United States (15):
  - Research Site, Phoenix, Arizona
  - Research Site, San Francisco, California
  - Research Site, New Haven, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Durham, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Seattle, Washington
- China (3):
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Italy (3):
  - Research Site, Benevento
  - Research Site, Milan
  - Research Site, Roma
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Osakasayama-shi
- Singapore (2):
  - Research Site, Bukit Merah
  - Research Site, Singapore
- South Korea (4):
  - Research Site, Busan
  - Research Site, Junggu
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Pamplona
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Kelley RK, Sangro B, Harris W, Ikeda M, Okusaka T, Kang YK, Qin S, Tai DW, Lim HY, Yau T, Yong WP, Cheng AL, Gasbarrini A, Damian S, Bruix J, Borad M, Bendell J, Kim TY, Standifer N, He P, Makowsky M, Negro A, Kudo M, Abou-Alfa GK. Safety, Efficacy, and Pharmacodynamics of Tremelimumab Plus Durvalumab for Patients With Unresectable Hepatocellular Carcinoma: Randomized Expansion of a Phase I/II Study. J Clin Oncol. 2021 Sep 20;39(27):2991-3001. doi: 10.1200/JCO.20.03555. Epub 2021 Jul 22. PMID 34292792
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4190C00022&attachmentIdentifier=0f980967-e716-4140-b0a7-995d874ae095&fileName=D4190C00022_SAP_edition_8-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4190C00022&attachmentIdentifier=37fea32a-6df6-405e-a3d1-24e72659273c&fileName=d4190c00022-exploratory-study-protocol-amendment-6-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4190C00022&attachmentIdentifier=b716d7b7-acde-479b-b4a3-a2c981f1902f&fileName=d4190c00022-CSR-synopsis-final-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results data are reported per the primary completion date (data cut-off date of 06Nov2020).
Groups:
- Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg: Participants in Part 1A (safety run-in cohort) and Part 1 B (efficacy-gating cohort) received tremelimumab 1 mg/kg every 4 weeks (Q4W) 4 doses and durvalumab 20 mg/kg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
- Parts 2 and 3: Durvalumab 1500 mg: Participants received durvalumab 1500 mg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
- Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg: Participants received tremelimumab 300 mg 1 dose and durvalumab 1500 mg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow, or development of other reason for treatment discontinuation, whichever occurred first.
- Parts 2 and 3: Tremelimumab 750 mg: Participants received tremelimumab 750 mg Q4W 7 doses followed by every 12 weeks (Q12W) until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
- Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg: Participants received tremelimumab 75 mg Q4W 4 doses and durvalumab 1500 mg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
- Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg: Participants received durvalumab 1120 mg and bevacizumab 15 mg/kg every 3 weeks (Q3W) until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
- China Cohort: Durvalumab 20 mg/kg: Participants received durvalumab 20 mg/kg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
- China Cohort: Tremelimumab 10 mg/kg: Participants received tremelimumab 10 mg/kg Q4W 7 doses followed by Q12W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
- China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg: Participants received tremelimumab 1 mg/kg Q4W 4 doses and durvalumab 20 mg/kg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
Period: Overall Study
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Started | 40 | 104 | 75 | 69 | 84 | 47 | 3 | 5 | 6
Treated | 40 | 101 | 74 | 69 | 82 | 47 | 3 | 5 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 40 | 104 | 75 | 69 | 84 | 47 | 3 | 5 | 6
Not completed — Death | 31 | 74 | 47 | 54 | 63 | 18 | 2 | 5 | 5
Not completed — Withdrawal by Subject | 4 | 7 | 4 | 3 | 3 | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Not completed — Other | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Ongoing at the time of data cut-off date | 5 | 20 | 23 | 12 | 15 | 26 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants (Parts 2A and 3) or participants who were allocated to treatment (Parts 1A, 1B, 2B, and 4), including participants who were randomized in error.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Total
Number analyzed (Participants) | 40 | 104 | 75 | 69 | 84 | 47 | 3 | 5 | 6 | 433
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 27 | 52 | 34 | 41 | 48 | 26 | 3 | 5 | 5 | 241
  >=65 to < 75 years | 8 | 33 | 31 | 18 | 26 | 13 | 0 | 0 | 1 | 130
  > 75 years | 5 | 19 | 10 | 10 | 10 | 8 | 0 | 0 | 0 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 10 | 12 | 14 | 6 | 1 | 0 | 0 | 65
  Male | 30 | 92 | 65 | 57 | 70 | 41 | 2 | 5 | 6 | 368
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 4 | 4 | 5 | 0 | 0 | 1 | 0 | 21
  Not Hispanic or Latino | 38 | 99 | 71 | 65 | 79 | 47 | 3 | 4 | 6 | 412
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Asian | 19 | 55 | 44 | 39 | 47 | 39 | 3 | 5 | 6 | 257
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 3 | 10 | 4 | 2 | 5 | 1 | 0 | 0 | 0 | 25
  White | 15 | 35 | 27 | 26 | 30 | 7 | 0 | 0 | 0 | 140
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as treatment-related toxicity that occurred during DLT evaluation period including: any Grade 4 immune-related adverse event (irAE), any Grade 3 colitis or any Grade 3 noninfectious pneumonitis irrespective of duration, any >= Grade 2 pneumonitis that does not resolve to <= Grade 1 within 7 days of initiation of maximal supportive care, any other Grade 3 irAE (excluding colitis or pneumonitis) that does not downgrade to Grade 2 within 7 days after onset of the event despite optimal medical management including systemic corticosteroids or does not downgrade to <= Grade 1 or baseline within 14 days, liver transaminase elevation > 8 × upper limit of normal (ULN) or total bilirubin > 5 × ULN, aspartate aminotransferase or alanine aminotransferase > 3 × ULN with concurrent increase in total bilirubin > 2 × ULN without evidence of cholestasis or alternative explanations, and any >= Grade 3 non-irAE (except for the protocol stated conditions).
Time Frame: From Day 1 to Day 28 after first dose of study drug
Population: DLT evaluable set included all Part 1A participants who received at least 1 dose of study drug and completed the safety follow-up through the DLT evaluation period (Days 1 to 28 after first dose of study drug) or experienced any DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1A: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg: Participants in Part 1A (safety run-in cohort) received tremelimumab 1 mg/kg every 4 weeks (Q4W) 4 doses and durvalumab 20 mg/kg Q4W until confirmed progressive disease, withdrawal of consent, lost to follow-up, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Part 1A: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 16
Participants | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: From Day 1 through the 12 months after the first dose of study drug given to the last participant enrolled in the study (approximately 61 months)
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 40 | 101 | 74 | 69 | 82 | 47 | 3 | 5 | 5
Participants
  Any TEAEs | 38 | 95 | 73 | 67 | 80 | 45 | 3 | 5 | 5
  Any TESAEs | 22 | 45 | 32 | 36 | 37 | 17 | 1 | 3 | 4

3. Primary Outcome: Number of Participants With Clinically Important Changes in Hematology and Clinical Chemistry Parameters
Description: Participants with clinically important Common Terminology Criteria for Adverse Events (CTCAE) grade changes to 3 or 4 in hematology and chemistry parameters are reported. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: Safety analysis set included all participants who received at least one dose of study drug. 'Number of participants analyzed' denotes only those participants for whom hematological and clinical chemistry parameter were analyzed. 'Number Analyzed' denotes the participants analyzed for the specified laboratory parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 39 | 100 | 74 | 68 | 81 | 46 | 3 | 5 | 4
Participants
  Hemoglobin: number analyzed (Participants) | 38 | 99 | 71 | 67 | 79 | 44 | 3 | 4 | 3
  Hemoglobin | 0 | 5 | 6 | 6 | 6 | 0 | 0 | 1 | 1
  Leukocytes: number analyzed (Participants) | 38 | 99 | 71 | 67 | 79 | 44 | 3 | 4 | 3
  Leukocytes | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
  Lymphocytes: number analyzed (Participants) | 29 | 75 | 52 | 55 | 65 | 24 | 3 | 4 | 3
  Lymphocytes | 3 | 7 | 10 | 4 | 8 | 2 | 0 | 1 | 0
  Neutrophils: number analyzed (Participants) | 33 | 75 | 51 | 55 | 65 | 32 | 3 | 4 | 3
  Neutrophils | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Platelets: number analyzed (Participants) | 37 | 99 | 71 | 67 | 79 | 44 | 3 | 4 | 3
  Platelets | 3 | 5 | 0 | 2 | 4 | 3 | 1 | 0 | 0
  Activated Partial Thromboplastin Time: number analyzed (Participants) | 34 | 98 | 69 | 68 | 78 | 44 | 3 | 4 | 3
  Activated Partial Thromboplastin Time | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Fibrinogen: number analyzed (Participants) | 34 | 95 | 66 | 64 | 76 | 44 | 3 | 4 | 3
  Fibrinogen | 5 | 5 | 5 | 2 | 5 | 3 | 0 | 0 | 0
  Prothrombin Intl. Normalized Ratio: number analyzed (Participants) | 39 | 100 | 74 | 67 | 81 | 46 | 3 | 5 | 4
  Prothrombin Intl. Normalized Ratio | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0
  Alanine Aminotransferase: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Alanine Aminotransferase | 3 | 7 | 13 | 5 | 10 | 1 | 0 | 0 | 0
  Albumin: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Albumin | 1 | 5 | 0 | 3 | 3 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Alkaline Phosphatase | 3 | 13 | 4 | 6 | 8 | 3 | 1 | 0 | 1
  Aspartate Aminotransferase: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Aspartate Aminotransferase | 5 | 25 | 19 | 16 | 17 | 4 | 0 | 1 | 1
  Bilirubin: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Bilirubin | 2 | 12 | 4 | 6 | 9 | 2 | 0 | 0 | 0
  Calcium - Hyper: number analyzed (Participants) | 37 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Calcium - Hyper | 0 | 4 | 0 | 1 | 3 | 1 | 0 | 0 | 0
  Calcium - Hypo: number analyzed (Participants) | 37 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Calcium - Hypo | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Creatinine: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Creatinine | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose - Hyper: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Glucose - Hyper | 4 | 8 | 14 | 6 | 5 | 2 | 0 | 0 | 0
  Glucose - Hypo: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Glucose - Hypo | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Magnesium - Hyper: number analyzed (Participants) | 37 | 98 | 70 | 67 | 78 | 45 | 3 | 4 | 3
  Magnesium - Hyper | 2 | 7 | 3 | 2 | 2 | 2 | 0 | 0 | 0
  Magnesium - Hypo: number analyzed (Participants) | 37 | 98 | 70 | 67 | 78 | 45 | 3 | 4 | 3
  Magnesium - Hypo | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Potassium - Hyper: number analyzed (Participants) | 38 | 98 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Potassium - Hyper | 4 | 4 | 2 | 0 | 3 | 1 | 0 | 0 | 0
  Potassium - Hypo: number analyzed (Participants) | 38 | 98 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Potassium - Hypo | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0
  Sodium - Hyper: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Sodium - Hyper | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium - Hypo: number analyzed (Participants) | 38 | 99 | 71 | 67 | 78 | 45 | 3 | 4 | 3
  Sodium - Hypo | 9 | 12 | 7 | 13 | 11 | 6 | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Vital sign assessment included pulse rate, blood pressure, temperature, weight, and respiratory rate. Vital signs abnormalities recorded as TEAEs are reported. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 40 | 101 | 74 | 69 | 82 | 47 | 3 | 5 | 5
Participants
  Hypertension | 1 | 4 | 4 | 2 | 3 | 6 | 0 | 0 | 0
  Hypotension | 0 | 4 | 0 | 3 | 2 | 0 | 0 | 0 | 0
  Systolic hypertension | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight decreased | 4 | 4 | 4 | 4 | 4 | 2 | 0 | 0 | 1
  Weight increased | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
  Palpitations | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Pyrexia | 6 | 6 | 14 | 9 | 14 | 4 | 2 | 2 | 1

5. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Reported as Treatment-Emergent Adverse Events
Description: Number of participants with ECG abnormalities recorded as TEAEs are reported. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 40 | 101 | 74 | 69 | 82 | 47 | 3 | 5 | 5
Participants
  Acute myocardial infarction | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Angina pectoris | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
  Angina unstable | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Atrial fibrillation | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 0
  Cardiac failure chronic | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac failure congestive | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Coronary artery disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sinus bradycardia | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Tachycardia | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Atrioventricular block first degree | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac arrest | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myocardial infarction | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

6. Secondary Outcome: Overall Objective Response Rate (ORR) Based on Investigator Assessments and Blinded Independent Central Review (BICR)
Description: Disease assessments based on investigator assessments and BICR review were determined by using Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1) guidelines. The ORR is defined as best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR). The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: Full analysis set included all randomized participants (Parts 2A and 3) or participants who were allocated to treatment (Parts 1, 2B, and 4), including participants who were randomized in error. Analysis of disease assessments based on BICR for Part 1 and China cohorts were not planned and hence not performed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 40 | 104 | 75 | 69 | 84 | 47 | 3 | 5 | 6
Percentage of participants
  ORR based on BICR: number analyzed (Participants) | 0 | 104 | 75 | 69 | 84 | 47 | 0 | 0 | 0
  ORR based on BICR |  | 11.5 [6.1 to 19.3] | 24.0 [14.9 to 35.3] | 7.2 [2.4 to 16.1] | 9.5 [4.2 to 17.9] | 21.3 [10.7 to 35.7] |  |  |
  ORR based on Investigator assessments | 20.0 [9.1 to 35.6] | 11.5 [6.1 to 19.3] | 21.3 [12.7 to 32.3] | 8.7 [3.3 to 18.0] | 8.3 [3.4 to 16.4] | 34.0 [20.9 to 49.3] | 33.3 [0.8 to 90.6] | NA [NA to NA] — No participants reported a best overall response of CR or PR. | NA [NA to NA] — No participants reported a best overall response of CR or PR.

7. Secondary Outcome: Disease Control Rate (DCR) Based on Investigator Assessments and BICR
Description: Disease assessments based on investigator assessments and BICR review were determined by using RECIST v1.1 guidelines. The DCR is defined as a BOR of confirmed CR, confirmed PR, or stable disease (SD). A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) that were separated by at least 4 weeks with no evidence of progression in-between. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 40 | 104 | 75 | 69 | 84 | 47 | 3 | 5 | 6
Percentage of participants
  DCR based on BICR: number analyzed (Participants) | 0 | 104 | 75 | 69 | 84 | 47 | 0 | 0 | 0
  DCR based on BICR |  | 37.5 | 45.3 | 49.3 | 36.9 | 55.3 |  |  |
  DCR based on Investigator assessments | 60.0 | 45.2 | 50.7 | 47.8 | 34.5 | 63.8 | 33.3 | 20.0 | 16.7

8. Secondary Outcome: Time to Response (TTR) Based on Investigator Assessments and BICR
Description: Disease assessments based on investigator assessments and BICR review were determined by using RECIST v1.1 guidelines. The TTR is defined as the time from randomization for Parts 2A and 3, and time from first dose for Parts 1, 2B, and 4 until the first documentation of a subsequently confirmed OR (confirmed CR or confirmed PR). A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) that were separated by at least 4 weeks with no evidence of progression in-between. The TTR was estimated using Kaplan-Meier method. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: Full analysis set included all randomized participants (Parts 2A and 3) or participants who were allocated to treatment (Parts 1, 2B, and 4), including participants who were randomized in error. Analysis of disease assessments based on BICR for Part 1 and China cohorts were not planned and hence not performed. The TTR was analyzed for participants who achieved OR per BICR and/or investigator assessments. 'Number Analyzed' denotes participants who achieved OR.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 8 | 12 | 18 | 6 | 8 | 16 | 1 | 0 | 0
Months
  TTR based on BICR: number analyzed (Participants) | 0 | 12 | 18 | 5 | 8 | 10 | 0 | 0 | 0
  TTR based on BICR |  | 3.65 [2.71 to 5.59] | 2.28 [1.81 to 3.68] | 1.81 [1.81 to 1.84] | 2.86 [1.84 to 3.83] | 2.10 [1.87 to 4.11] |  |  |
  TTR based on Investigator assessments: number analyzed (Participants) | 8 | 12 | 16 | 6 | 7 | 16 | 1 | 0 | 0
  TTR based on Investigator assessments | 2.68 [1.82 to 4.60] | 3.68 [1.81 to 5.55] | 1.86 [1.77 to 5.59] | 2.74 [1.81 to 5.32] | 3.88 [1.81 to 5.32] | 2.10 [1.94 to 4.12] | 5.55 [5.55 to 5.55] |  |

9. Secondary Outcome: Duration of Response (DoR) Based on Investigator Assessments and BICR
Description: The DoR is defined as the time from the date of first documented OR (confirmed CR or confirmed PR) until date of documented progression (PD) based on investigator assessments and BICR review by using RECIST v1.1 or death in absence of disease progression. A confirmed CR is defined in above outcome measures. The PD is defined at least 20% increase in sum of diameters of target lesions (compared with nadir at 2 consecutive visits with an absolute increase of 5 mm), unequivocal progression of existing non-target lesions or new lesion. For participants who were alive and no documented PD at the time of data cutoff for analysis, DoR was censored at the last evaluable disease assessment date. The DoR was estimated using Kaplan-Meier method. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: Full analysis set included all randomized participants (Parts 2A and 3) or participants who were allocated to treatment (Parts 1, 2B, and 4), including participants who were randomized in error. Analysis of disease assessments based on BICR for Part 1 and China cohorts were not planned and hence not performed. The DoR was analyzed for participants who achieved OR per BICR and/or investigator assessments. 'Number Analyzed' denotes participants who achieved OR.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 8 | 12 | 18 | 6 | 8 | 16 | 1 | 0 | 0
Months
  DoR based on BICR: number analyzed (Participants) | 0 | 12 | 18 | 5 | 8 | 10 | 0 | 0 | 0
  DoR based on BICR |  | 14.95 [8.54 to NA] — 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | 18.43 [5.59 to 23.95] | 23.95 [4.07 to NA] — 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | 13.21 [10.15 to NA] — 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | NA [6.28 to NA] — Median and 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. |  |  |
  DoR based on Investigator assessments: number analyzed (Participants) | 8 | 12 | 16 | 6 | 7 | 16 | 1 | 0 | 0
  DoR based on Investigator assessments | 16.66 [8.41 to NA] — 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | NA [19.02 to NA] — Median and 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | 23.95 [5.59 to NA] — 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | 27.53 [27.53 to NA] — 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | 13.21 [12.85 to NA] — 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | 10.51 [10.51 to NA] — 75th percentile could not be derived due to insufficient events being observed at the time of the analysis. | 7.39 [7.39 to 7.39] |  |

10. Secondary Outcome: Time to Progression (TTP) Based on Investigator Assessments and BICR
Description: Disease assessments based on investigator assessments and BICR review were determined by using RECIST v1.1 guidelines. The TTP was defined as the time from randomization for Parts 2A and 3, and time from first dose for Parts 1, 2B, and 4 to the first documentation of radiographic disease progression. However, if the participant died without tumor progression, they were censored at the time of death. Participants with no documented PD by the data cutoff date for TTP analysis were censored at the date of their last evaluable disease assessment. The TTP was estimated using Kaplan-Meier method. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 40 | 104 | 75 | 69 | 84 | 47 | 3 | 5 | 6
Months
  TTP based on BICR: number analyzed (Participants) | 0 | 104 | 75 | 69 | 84 | 47 | 0 | 0 | 0
  TTP based on BICR |  | 2.10 [1.87 to 3.52] | 3.71 [1.91 to 5.55] | 2.76 [1.87 to 5.42] | 1.87 [1.81 to 3.48] | 4.30 [2.10 to 6.24] |  |  |
  TTP based on Investigator assessments | 3.68 [2.23 to 6.77] | 3.38 [2.00 to 4.67] | 3.68 [2.07 to 5.52] | 2.60 [1.87 to 5.29] | 1.87 [1.77 to 3.48] | 7.46 [4.01 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 1.81 [1.64 to 12.91] | 3.75 [1.81 to 3.75] | 2.68 [1.84 to 3.48]

11. Secondary Outcome: Progression Free Survival (PFS) Based on Investigator Assessments and BICR
Description: Disease assessments based on investigator assessments and BICR review were determined by using RECIST v1.1 guidelines. The PFS is defined as the time from randomization for Parts 2A and 3, and time from first dose for Parts 1, 2B, and 4 until the first documentation of radiographic disease progression or death due to any cause, whichever occurs first. The PD is defined at least 20% increase in the sum of diameters of target lesions (compared with the nadir at 2 consecutive visits with an absolute increase of 5 mm), unequivocal progression of existing non-target lesions or new lesion. Participants who were alive with no documented PD by the data cutoff date for PFS analysis were censored at the date of their last evaluable disease assessment. The PFS was estimated using Kaplan-Meier method. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 40 | 104 | 75 | 69 | 84 | 47 | 3 | 5 | 6
Months
  PFS based on BICR: number analyzed (Participants) | 0 | 104 | 75 | 69 | 84 | 47 | 0 | 0 | 0
  PFS based on BICR |  | 2.07 [1.84 to 2.86] | 2.17 [1.91 to 5.42] | 2.69 [1.87 to 5.29] | 1.87 [1.77 to 2.53] | 4.17 [2.10 to 6.24] |  |  |
  PFS based on Investigator assessments | 3.52 [1.87 to 5.29] | 2.40 [1.91 to 3.65] | 3.52 [2.07 to 5.42] | 2.60 [1.87 to 3.71] | 1.81 [1.77 to 2.40] | 6.24 [3.94 to 12.55] | 1.81 [1.64 to 12.91] | 2.20 [1.81 to 3.75] | 1.87 [0.66 to 3.48]

12. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from randomization for Parts 2A and 3, and time from first dose for Parts 1, 2B, and 4 until death due to any cause. If there was no death reported for a participant by the data cut-off date for overall survival analysis, OS was censored at the last known alive date. The OS was estimated using Kaplan-Meier method. There will be no updated results for this outcome measure at the time of end of study.
Time Frame: as for outcome 2
Population: Full analysis set included all randomized participants (Parts 2A and 3) or participants who were allocated to treatment (Parts 1, 2B, and 4), including participants who were randomized in error.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
Number analyzed (Participants) | 40 | 104 | 75 | 69 | 84 | 47 | 3 | 5 | 6
Months | 12.58 [6.87 to 20.99] | 12.91 [8.74 to 16.79] | 17.05 [10.55 to 22.83] | 17.05 [11.33 to 20.24] | 11.30 [8.38 to 14.95] | NA [12.52 to NA] — Median and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 30.69 [13.96 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 3.52 [2.20 to 20.96] | 6.28 [0.66 to 23.82]

ADVERSE EVENTS:
Time Frame: From Day 1 through the 12 months after the first dose of study drug given to the last participant enrolled in the study (approximately 61 months)
Description: All-Cause Mortality was evaluated per 'Full analysis set' which included all randomized participants (Parts 2A and 3) or participants who were allocated to treatment (Parts 1, 2B, and 4), including participants who were randomized in error.
  The AE data was evaluated per 'Safety population' which included all participants who received at least one dose of study drug.
Arm/Group | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg | Parts 2 and 3: Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg | Parts 2 and 3: Tremelimumab 750 mg | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg | China Cohort: Durvalumab 20 mg/kg | China Cohort: Tremelimumab 10 mg/kg | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 31/40 | 78/104 | 49/75 | 55/69 | 64/84 | 18/47 | 2/3 | 5/5 | 5/6
Serious Adverse Events (participants affected / at risk) | 22/40 | 45/101 | 32/74 | 36/69 | 37/82 | 17/47 | 1/3 | 3/5 | 4/5
Other Adverse Events (participants affected / at risk) | 37/40 | 92/101 | 73/74 | 66/69 | 80/82 | 45/47 | 3/3 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg (N=40) | Parts 2 and 3: Durvalumab 1500 mg (N=101) | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg (N=74) | Parts 2 and 3: Tremelimumab 750 mg (N=69) | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg (N=82) | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg (N=47) | China Cohort: Durvalumab 20 mg/kg (N=3) | China Cohort: Tremelimumab 10 mg/kg (N=5) | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg (N=5)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (5) | 3 (3) | 0 (0) | 0 (0) | 2 (9) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipogranuloma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 9 (10) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Listeria sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Listeriosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperammonaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg (N=40) | Parts 2 and 3: Durvalumab 1500 mg (N=101) | Parts 2 and 3: Tremelimumab 300 mg + Durvalumab 1500 mg (N=74) | Parts 2 and 3: Tremelimumab 750 mg (N=69) | Parts 2 and 3: Tremelimumab 75 mg + Durvalumab 1500 mg (N=82) | Part 4: Durvalumab 1120 mg + Bevacizumab 15 mg/kg (N=47) | China Cohort: Durvalumab 20 mg/kg (N=3) | China Cohort: Tremelimumab 10 mg/kg (N=5) | China Cohort: Tremelimumab 1 mg/kg + Durvalumab 20 mg/kg (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 7 (12) | 10 (13) | 9 (16) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 2 (2) | 0 (0) | 4 (6) | 2 (2) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 2 (2) | 6 (6) | 1 (1) | 4 (7) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 12 (13) | 8 (8) | 4 (4) | 8 (11) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Immune-mediated endocrinopathy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 10 (10) | 8 (8) | 6 (6) | 5 (7) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 15 (17) | 10 (12) | 15 (19) | 11 (13) | 7 (8) | 0 (0) | 1 (1) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 5 (5) | 3 (3) | 6 (6) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 6 (6) | 8 (8) | 10 (11) | 6 (7) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (7) | 12 (14) | 8 (10) | 7 (8) | 10 (12) | 5 (7) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 14 (17) | 17 (20) | 14 (20) | 19 (29) | 14 (23) | 9 (10) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal varices (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysbiosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 12 (14) | 10 (10) | 14 (15) | 11 (11) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation lip (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (5) | 7 (7) | 4 (4) | 8 (10) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 13 (14) | 23 (28) | 17 (20) | 19 (22) | 15 (19) | 10 (13) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal hyperaemia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 15 (15) | 12 (14) | 5 (6) | 12 (13) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (6) | 4 (6) | 11 (20) | 9 (12) | 11 (15) | 3 (4) | 2 (2) | 2 (2) | 1 (3)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 3 (5) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis b (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (5) | 3 (3) | 8 (9) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 7 (8) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired pigmented retinopathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (3) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (11) | 23 (33) | 17 (28) | 11 (19) | 15 (19) | 2 (2) | 3 (7) | 2 (2) | 2 (3)
Ammonia increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 4 (5) | 8 (9) | 12 (20) | 8 (10) | 8 (12) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 9 (12) | 26 (33) | 23 (38) | 19 (29) | 21 (27) | 6 (7) | 3 (6) | 3 (3) | 2 (3)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 11 (18) | 7 (7) | 7 (10) | 6 (8) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 10 (14) | 7 (11) | 10 (16) | 7 (7) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 2 (3) | 7 (12) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 6 (8) | 5 (5) | 6 (11) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Granulocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis b dna increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 4 (4) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 7 (9) | 5 (7) | 12 (20) | 14 (30) | 6 (10) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 4 (6) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 6 (13) | 2 (5) | 5 (7) | 2 (9) | 5 (9) | 1 (5) | 0 (0) | 1 (3)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroxine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 4 (4) | 4 (4) | 4 (5) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (7) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 14 (15) | 10 (11) | 16 (16) | 14 (17) | 12 (14) | 0 (0) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 2 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 8 (11) | 7 (8) | 4 (8) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 2 (6) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 7 (10) | 3 (3) | 4 (5) | 4 (5) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoferritinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4) | 6 (7) | 5 (6) | 3 (3) | 4 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (9) | 4 (4) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 5 (7) | 2 (2) | 5 (9) | 5 (6) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (9) | 8 (9) | 9 (10) | 7 (8) | 5 (9) | 0 (0) | 0 (0) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 15 (16) | 2 (2) | 6 (7) | 6 (6) | 6 (8) | 1 (1) | 0 (0) | 0 (0)
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (6) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 4 (4) | 2 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (7) | 6 (6) | 1 (1) | 6 (6) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 8 (9) | 2 (2) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 7 (7) | 2 (2) | 8 (8) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 11 (17) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 12 (12) | 15 (17) | 11 (17) | 15 (18) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (10) | 4 (5) | 5 (5) | 6 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12) | 20 (26) | 29 (42) | 28 (38) | 21 (25) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura senile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 13 (13) | 27 (33) | 20 (27) | 14 (15) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 8 (10) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloody discharge (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 4 (6) | 4 (5) | 2 (2) | 3 (9) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inferior vena caval occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT02519348/Prot_004.pdf
  • Statistical Analysis Plan (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT02519348/SAP_005.pdf